CLINICAL TRIAL: NCT05107505
Title: Evaluation of The Factors Affecting Bowel Preparation Adequacy for Colonoscopy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Alexandra Hospital, Athens, Greece (Other)
Responsible Party: Principal Investigator, SPYRIDON MICHOPOULOS, Head Of The Gastroenterology Departement, Alexandra Hospital, Athens, Greece
Other Study IDs: Alexandra Bowel Preparation
Record Dates: First submitted 2021-10-26; First posted 2021-11-04 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Bowel Preparation; Preparation for Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A prospective observational study in order to:

1. st: Identify epidemiological, clinical, and preparation-related factors that can predict improper preparation leading to better management of the patients with non adequate preparation.
2. nd: Evaluation of the effect of the time of preparation and endoscopy initiation time on the outcome of intestinal preparation for colonoscopy.

DETAILED DESCRIPTION:
Unsuccessful preparation for lower gastrointestinal endoscopy is to date the main obstacle to a comprehensive examination and the main reason for its recurrence. It is also directly related to its diagnostic value.

The literature shows that the diet prior to colonoscopy, the time of assumption of the preparation and certain epidemiological and clinical characteristics of the patient can affect the outcome of the intestinal preparation for colonoscopy.

This seems that adequasy of colonoscopy affects a number of qualitative indicators of lower gastrointestinal endoscopy, such as the duration, the catheterization of the fundus of the cecum and the number of polyps found.

This is a prospective observational study in order to:

1. st: Identify epidemiological, clinical, and preparation-related factors that can predict improper preparation leading to better management of the patients with non adequate preparation.
2. nd: Evaluation of the effect of the time of preparation and endoscopy initiation time on the outcome of intestinal preparation for colonoscopy.

With starting date:01/07/2021 and expiration date:30/06/2022 (duration: 12 months). All patients who come to the Gastroenterology Department of Alexandra Hospital for endoscopy of the lower digestive tract are eligible for the research protocol. Patients younger than 18 years old or patients who refuse to participate are excluded.

The study has 3 phases. Phase 0 entails the completion of a questionnaire that will include epidemiological, clinical and preparation-related data in all patients who undergoing colonoscopy at the Endoscopy Department. Phase I incorporates Completion of data related to the time of the examination, the result of the preparation (Boston Bowel Preparation Scale) as well as the findings of the endoscopic examination and phase II includes the statistical analysis of the data.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing colonoscopy:

* Age > 18 years
* Have been prepared for lower gastrointestinal endoscopy
* Have agreed to participate in the study

Exclusion Criteria:

* Age <18 years
* Non-acceptance of participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1000 adult patients undergoing colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-07-14 (Estimated); Study Completion 2023-07-14 (Estimated)

PRIMARY OUTCOMES:
improper bowel preparation | 01/07/2021-30/06/2022
  Identify epidemiological, clinical, and preparation-related factors that can predict improper preparation leading to better management of the patients with non adequate preparation.

SECONDARY OUTCOMES:
quality of preparation for colonoscopy | 01/07/2021-30/06/2022
  Evaluation of the effect of the time of preparation and endoscopy initiation time on the outcome of intestinal preparation for colonoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandra General Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lai EJ, Calderwood AH, Doros G, Fix OK, Jacobson BC. The Boston bowel preparation scale: a valid and reliable instrument for colonoscopy-oriented research. Gastrointest Endosc. 2009 Mar;69(3 Pt 2):620-5. doi: 10.1016/j.gie.2008.05.057. Epub 2009 Jan 10. PMID 19136102
- [Background] Hassan C, Bretthauer M, Kaminski MF, Polkowski M, Rembacken B, Saunders B, Benamouzig R, Holme O, Green S, Kuiper T, Marmo R, Omar M, Petruzziello L, Spada C, Zullo A, Dumonceau JM; European Society of Gastrointestinal Endoscopy. Bowel preparation for colonoscopy: European Society of Gastrointestinal Endoscopy (ESGE) guideline. Endoscopy. 2013;45(2):142-50. doi: 10.1055/s-0032-1326186. Epub 2013 Jan 18. PMID 23335011
- [Background] Millien VO, Mansour NM. Bowel Preparation for Colonoscopy in 2020: A Look at the Past, Present, and Future. Curr Gastroenterol Rep. 2020 May 6;22(6):28. doi: 10.1007/s11894-020-00764-4. PMID 32377915